CLINICAL TRIAL: NCT02579278
Title: Circulating Tumour DNA (ctDNA) in Patients With Colorectal Cancer and the Relationship to Imaging Features of Extramural Venous Invasion
Acronym: ctDNA
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: DOCUMAS: 23HH8182
Record Dates: First submitted 2015-10-06; First posted 2015-10-19 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Rectal Cancer
Keywords: EMVI; Extramural Venous Invasion; mrEMVI; Rectal Cancer; ctDNA; Neoplasm DNA; MRI
MeSH Terms: conditions — Neoplasms; Rectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each patient will have two blood samples taken that will be analysed for ctDNA. One blood sample will be taken at the time of preoperative assessment, after chemoradiotherapy, and a further sample will be taken intraoperatively, from the peripheral vein of the patient's arm. For each of the blood samples the presence or absence of ctDNA mutations (kras and p53) will be identified.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- mrEMVI positive rectal tumours: Patients will be registered whose rectal tumours are mrEMVI positive (i.e. EMVI is present in baseline and post-chemoradiotherapy MRI scans).
  Interventions: Other: Blood sample (mrEMVI positive patient)
- mrEMVI negative rectal tumours: Patients registered who were mrEMVI positive at baseline MRI but have become mrEMVI negative post-chemoradiotherapy.
  Interventions: Other: Blood sample (mrEMVI negative patient)

INTERVENTIONS:
Other: Blood sample (mrEMVI positive patient) — Two blood samples are taken from each patient with mrEMVI positive tumours post chemoradiotherapy. One pre-surgery and one during surgery from a peripheral vein.
  Groups: mrEMVI positive rectal tumours
Other: Blood sample (mrEMVI negative patient)
  Other Names: Two blood samples are taken from each patient with mrEMVI negative tumours post chemoradiotherapy. One pre-surgery and one during surgery from a peripheral vein.
  Groups: mrEMVI negative rectal tumours

SUMMARY:
This study does not involve randomization or treatment. Eligible patients have colorectal adenocarcinoma with no metastases eligible for curative surgery. A pre operative staging scan must have been completed within 6 weeks prior to surgery. Two x 20ml blood samples will be taken from each patient, one prior to and one during or within 24hrs after surgery. Patients are annually followed up to 3 years.

DETAILED DESCRIPTION:
A multicentre observational study, ctDNA aims to provide the evidence base for metatstatic disease being caused by vascular methods of spread by determining if there is a link between EMVI status and ctDNA

ELIGIBILITY:
Inclusion Criteria:

1. Have a biopsy-confirmed colorectal adenocarcinoma
2. Is eligible for curative surgery
3. Has no metastatic disease on CT scan
4. Has completed pre-operative staging scan within six weeks prior to surgery
5. Have provided written informed consent to participate in the study
6. Be aged 16 years or over

Exclusion Criteria:

1. Have metastatic disease (including resectable liver metastases)
2. Have a synchronous second malignancy
3. Are contraindicated for any imaging able to determine EMVI status

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 adult patients presenting with primary colorectal cancer proven on biopsy with no evidence of metastatic disease on CT and who are eligible for curative surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
To determine if there is a link between EMVI status and ctDNA | Up to 2 years
  Proportion of patients who are EMVI positive demonstrating higher % mutation frequency of circulating cell-free and tumour specific DNA compared with patients who are EMVI negative.

SECONDARY OUTCOMES:
To investigate whether ctDNA levels change during surgery according to EMVI status | Up to 2 years
  Measure the intraoperative % mutation frequency of ctDNA in EMVI positive compared with EMVI negative patients
To investigate the effect of ctDNA status on patient survival outcomes | At 1, 2 and 3 years
  Record survival outcomes of patients who are: EMVI negative with low ctDNA levels, EMVI negative with high ctDNA levels, EMVI positive with low ctDNA levels, EMVI positive with high ctDNA levels

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, MD, Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - Queen Elizabeth the Queen Mother Hospital, Margate, Kent
  - St Mary's Hospital (Imperial), Hammersmith, London
  - Royal Marsden Hospital NHS Foundation Trust, Sutton, Surrey